CLINICAL TRIAL: NCT07258264
Title: Programa Educativo y Formativo Basado en la Entrevista Motivacional Para Pacientes Con SAHS en Tratamiento Con CPAP: MEntA
Brief Title: MEntA Program Based on Motivational Interview to Improve Adherence to Treatment of Obstructive Sleep Apnea With Continuous Positive Airway Pressure (CPAP)
Acronym: MEntA Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Air Liquide Healthcare Spain (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 3687
Record Dates: First submitted 2025-09-26; First posted 2025-12-02 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Apnea (Central and Obstructive)
MeSH Terms: conditions — Apnea | interventions — Motivational Interviewing

STUDY DESIGN:
Intervention Model Description: A randomized, controlled, single-centre trial design was performed
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Competency-based learning - Control (Active Comparator): Standard of Care Group: subjects undergoing this training intervention follow the standard procedure. It consists of a CPAP School for the initiation of therapy, and follow-up visits (in person and/or by telephone) that follow the frequencies indicated by the Spanish Society of Pulmonology and Thoracic Surgery (SEPAR). The CPAP School consists of a single session lasting around 80 minutes. The theoretical training includes the importance of adherence, as well as handling the equipment and accessories, cleaning and maintenance of the equipment, and prevention of complications and possible side effects. The practical training consists of showing patients how to carry out the technique themselves.
  Interventions: Behavioral: Competency-based learning
- Motivational Interviewing - MEntA (Experimental): subjects in this group underwent an intervention based on the motivational interviewing (MI) technique in CPAP School format for the initiation of therapy, and follow-up as indicated by SEPAR. MEntA CPAP School intervention consists of one session lasting approximately 90 minutes, which is divided into two blocks: educational activity and training activity. In the first block, an expert explains the concepts of sleep apnoea and the symptoms, while a patient shows the CPAP treatment and how to optimize this to the fullest. This block was reinforced with documentation in hard copy and digital format. The second block on training activity was based on working with the treatment, equipment, safety, hygiene and advice. MEntA has the specific contents but the key is in how these contents are treated with the patients, using the MI to the treatment of OSA with CPAP.
  Interventions: Behavioral: Motivational Interviewing (MI)

INTERVENTIONS:
Behavioral: Motivational Interviewing (MI) — Collaborative and person-centered counseling style designed to help people explore and resolve their ambivalence about change, thereby strengthening their intrinsic motivation to make positive behavioral changes
  Arms: Motivational Interviewing - MEntA
Behavioral: Competency-based learning — Consists of exposing the contents in a "classroom" format and promoting the acquisition of the contents of each aspect through practice. The training focuses on the skills of handling and use of CPAP
  Arms: Competency-based learning - Control

SUMMARY:
A randomized, controlled, single-centre trial design was performed. The interventions were standard of care vs MEntA Program based on motivational interview for adherence. The main outcome was the adherence with the CPAP therapy after 90 days of treatment. Secondary outcomes were the motivation, perceived competence, quality of life, sleepiness, emotional state, activities and social relations.

DETAILED DESCRIPTION:
The subjects enrolled in the study were required to have a diagnosis of OSA confirmed by polysomnography (PSG), be recommended for treatment with CPAP and be naïve to this type of intervention. The study excluded subjects requiring bi-level ventilation, such as those with central sleep apnoea syndrome, a CPAP assessment study, those with severe chronic obstructive pulmonary disease (COPD), cognitive disorders and those unable to understand the consent form to participate. Prior to enrolment in the study, all patients were informed in detail about the study and signed the consent form to participate. Standard of Care Group: subjects undergoing this training intervention follow the standard procedure. It consists of a CPAP School for the initiation of therapy, and follow-up visits (in person and/or by telephone) that follow the frequencies indicated by the Spanish Society of Pulmonology and Thoracic Surgery (SEPAR). The CPAP School consists of a single session lasting around 80 minutes. The theoretical training includes the importance of adherence, as well as handling the equipment and accessories, cleaning and maintenance of the equipment, and prevention of complications and possible side effects. The practical training consists of showing patients how to carry out the technique themselves.

MEntA Group: subjects in this group underwent an intervention based on the motivational interviewing (MI) technique in CPAP School format for the initiation of therapy, and follow-up as indicated by SEPAR. MEntA CPAP School intervention consists of one session lasting approximately 90 minutes, which is divided into two blocks: educational activity and training activity. In the first block, an expert explains the concepts of sleep apnoea and the symptoms, while a patient shows the CPAP treatment and how to optimize this to the fullest. This block was reinforced with documentation in hard copy and digital format. The second block on training activity was based on working with the treatment, equipment, safety, hygiene and advice. MEntA has the specific contents but the key is in how these contents are treated with the patients, using the MI to the treatment of OSA with CPAP.

For perceived competence was used the validated Questionnaire of Evaluation of Perceived Competence in Adherence to CPAP in OSA (CEPCA)9. This questionnaire consists of 3 categories and 13 items: knowledge of OSA and its associated risk; expectations regarding CPAP treatment; and confidence in overcoming obstacles associated with the use of this type of treatment. The scores obtained in the CEPCA imply they are positively related to quality of life and motivation and negatively related to daytime sleepiness.

The quality of life was assessed using the Visual Analogical Well-being Scale for apnoea10 and sleepiness was assessed using the Epworth Sleepiness Scale (ESS)11,12. Finally, emotional state, daily activities and social relationships were also measured using the following ad hoc question "Taking into account your sleep problems, how would say you are in terms of mood / activities / social relationships?". The answer alternatives are: Good, Normal / no change, Bad.

ELIGIBILITY:
Inclusion Criteria:

* To have a diagnosis of OSA confirmed by polysomnography (PSG)
* CPAP treatment prescription
* First time with this type of intervention.

Exclusion Criteria:

* Subjects requiring bi-level ventilation
* Pacients with central sleep apnoea syndrome
* Patients with severe chronic obstructive pulmonary disease (COPD)
* Patients with cognitive disorders and those unable to understand the consent form to participate.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2019-05-30 (Actual); Primary Completion 2019-10-21 (Actual); Study Completion 2019-10-21 (Actual)

PRIMARY OUTCOMES:
Adherence | From enrollment to the end of treatment at 90 days.
  Total number of night-time hours registered by the CPAP device

SECONDARY OUTCOMES:
Motivation for the use of CPAP treatment. | Baseline, 30 days and 90 days
  Set of factors, both internal and external, that drive a person to initiate, maintain, and direct their behavior toward the use of CPAP. The Motivation to Use CPAP Scale (MUC-S) is used for its evaluation. It is a 5-point Likert-type scale from strongly agree (5) to strongly disagree (1). The possible range for the scale is 9-45. A higher score indicates greater motivation to use CPAP treatment.
Perceived competence | Baseline, 30 days and 90 days
  An individual's subjective belief in their own effectiveness and ability to learn and execute skills within a specific context, such as academics or social interactions. The OSA-CPAP Perceived Competence Evaluation Interview, composed of 13 items with a Yes or No response option, is used for its evaluation. Minimum score = 0; Maximum score = 13. The higher the score, the more competent the patient perceives himself to be in the use of CPAP and the better his self-efficacy.
Well-being | Baseline, 30 days and 90 days.
  Subjective perception of a person about their overall well-being. For its evaluation, Visual analogical well-being scale for sleep apnea is used. It consists of a 120-mm straight line on which the patient indicates his or her health status with respect to the symptoms which were the motivation for the consultation (e.g., OSA). The ends of the line indicate the least favorable and the most favorable well-being status. It functions as an Analog Rating Scale, with scores ranging from 0 (minimum) to 10 (maximum). The higher the score, the better the well-being in relation to the symptoms of obstructive sleep apnea.
Sleepiness | Baseline, 30 days and 90 days
  Strong desire to sleep or a state of excessive drowsiness. For its evaluation, the Epworth test is used, a self-administered questionnaire with eight questions used to measure a person's general level of daytime sleepiness. It assesses the likelihood of dozing off in common situations, and a total score is calculated from (0) (never doze) to (3) (high chance of dozing) for each question. Minimum score = 0 and maximum score = 24. Scores between 0-10 are considered normal; scores between 11-14 are considered mild daytime sleepiness; scores between 15-18 are considered moderate daytime sleepiness; scores between 19-24 are considered severe daytime sleepiness.
Emotional state | Baseline, day 30 and day 90.
  Individual's experience of feelings and moods, such as happiness, sadness, anger, or anxiety, which can be influenced by internal factors and external events. For its evaluation, an ad hoc scale with 3 possible categories is used, which the patient chooses: bad (score 0), normal (score 1), better (score 2). A higher score is interpreted as a better mood
Daily activities | Baseline, Day 30 and Day 90
  Regular actions people perform each day, encompassing personal care (like bathing and eating), work or school, and leisure (like reading or hobbies). For its evaluation, an ad hoc scale with 3 possible categories is used, which the patient chooses: bad (score 0), normal (score 1), better (score 2). A higher score is interpreted as a greater ability to perform activities of daily living.
Social relationships | Baseline, Day 30 and Day 90
  Regular actions people perform each day, encompassing personal care (like bathing and eating), work or school, and leisure (like reading or hobbies). For its evaluation, an ad hoc scale with 3 possible categories is used, which the patient chooses: bad (score 0), normal (score 1), better (score 2). A higher score is interpreted as a greater ability to participate in social activities.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universitario de La Princesa, Madrid, Madrid, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Rudilla D, Landete P, Zamora E, Roman A, Vergara I, Ancochea J. MEntA Program Based on Motivational Interview to Improve Adherence to Treatment of Obstructive Sleep Apnea With Continuous Positive Airway Pressure (CPAP): A Randomized Controlled Trial. Open Respir Arch. 2021 Mar 16;3(2):100088. doi: 10.1016/j.opresp.2021.100088. eCollection 2021 Apr-Jun. PMID 37497068